CLINICAL TRIAL: NCT00960115
Title: Combined Phase I/II Clinical Study of EMD531444(L-BLP25 or BLP25 Liposome Vaccine) in Subjects With Stage III Unresectable Non-small Cell Lung Cancer Following Primary Chemoradiotherapy
Brief Title: Study of Tecemotide (L-BLP25) in Participants With Stage III Unresectable Non-small Cell Lung Cancer (NSCLC) Following Primary Chemoradiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR063325_009
Record Dates: First submitted 2009-08-05; First posted 2009-08-17 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Stage III; EMD531444; L-BLP25; Cyclophosphamide; Immunotherapy; Tecemotide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Single Person; Cyclophosphamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tecemotide (L-BLP25) + Cyclophosphamide (Experimental): Active
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Single low dose cyclophosphamide
- Placebo + Saline (Placebo Comparator): Control
  Interventions: Biological: Placebo; Other: Saline

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — After receiving a single low-dose cyclophosphamide, participants will receive weekly subcutaneous vaccinations with tecemotide (L-BLP25) (930 microgram [mcg]) for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with tecemotide (L-BLP25) (930 mcg) will be administered every 6 weeks until progressive disease (PD).
  Other Names: EMD531444; L-BLP25; BLP25 Liposome Vaccine
  Arms: Tecemotide (L-BLP25) + Cyclophosphamide
Drug: Single low dose cyclophosphamide — A single intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg/m^2) of cyclophosphamide will be administered 3 days prior to tecemotide (L-BLP25), the first vaccine treatment.
  Arms: Tecemotide (L-BLP25) + Cyclophosphamide
Biological: Placebo — After receiving single dose of saline, participants will receive weekly subcutaneous vaccinations with placebo that matches with tecemotide (L-BLP25) for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with placebo will be administered every 6 weeks until PD.
  Arms: Placebo + Saline
Other: Saline — A single dose of saline (sodium chloride, 9 grams per liter [g/L]) will be administered intravenously, 3 days prior to the start of placebo.
  Arms: Placebo + Saline

SUMMARY:
This is a phase I/II study in Japan to evaluate the safety of EMD531444 and its effects on survival time in patients with stage III unresectable non-small cell lung cancer.

DETAILED DESCRIPTION:
Phase I part is designed to evaluate the safety of EMD531444 930 microgram (mcg) dose to be used in phase II. Phase II part is designed to be conducted as randomized, double blind, placebo controlled study to compare overall survival time in all randomized subjects.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of concomitant or sequential chemoradiotherapy, consisting of a minimum of two cycles of platinum-based chemotherapy and a minimum radiation dose of greater than or equal to (>=) 50 Gray (Gy). Participant must have completed the primary thoracic chemoradiotherapy at least 4 weeks and no later than 12 weeks prior to randomization
* Written informed consent given before any study-related activities are carried out.
* Histologically or cytologically documented unresectable stage III NSCLC. Cancer stage must be confirmed and documented by Computed Tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) scan
* Documented stable disease or objective response, according to RECIST, after primary chemoradiotherapy for unresectable stage III disease, within four weeks prior to randomization
* Receipt of concomitant or sequential chemoradiotherapy, consisting of a minimum of two cycles of platinum-based chemotherapy and a minimum radiation dose of >= 50 Gy
* Eastern cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow function
* Greater than or equal to 20 years of age

Exclusion Criteria:

* Lung cancer-specific therapy (including surgery), other than primary chemoradiotherapy. Note: exploratory surgery before study entry is allowed
* Immunotherapy (e.g., interferons, tumor necrosis factor [TNF], interleukins, or biological response modifiers [granulocyte macrophage colony stimulating factor {GM-CSF}, granulocyte colony stimulating factor {G-CSF}, macrophage-colony stimulating factor {M-CSF}], monoclonal antibodies) received within four weeks prior to randomization
* Malignant pleural/pericardial effusion or pleural dissemination or separate tumor nodules in the same lobe at initial diagnosis and/or at study entry
* Past or current history of neoplasm other than lung carcinoma, except for adequately treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least five years
* Autoimmune disease
* A recognized immunodeficiency disease including cellular immunodeficiencies, hypogamma-globulinemia, or dysgammaglobulinemia; participants who have hereditary or congenital/acquired immunodeficiencies
* Any preexisting medical condition requiring chronic steroid or immunosuppressive therapy, including presence of diffuse radiation pneumonitis spreading out of the involved field
* Known Hepatitis B and/or C
* Clinically significant hepatic dysfunction
* Clinically significant renal dysfunction
* Clinically significant cardiac disease
* Splenectomy
* Infectious process that, in the opinion of the investigator, could compromise the subject's ability to mount an immune response
* Pregnant or breast-feeding women. Participants whom the investigator considers may be at risk of pregnancy will have a pregnancy test performed per institutional standard. Male and female subjects who have a reproductive ability, unless using effective contraception as determined by the investigator throughout the study until at least 6 months after the last study treatment
* Known drug abuse or alcohol abuse
* Legal incapacity or limited legal capacity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-12; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] Zhu J, Yuan Y, Wan X, Yin D, Li R, Chen W, Suo C, Song H. Immunotherapy (excluding checkpoint inhibitors) for stage I to III non-small cell lung cancer treated with surgery or radiotherapy with curative intent. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD011300. doi: 10.1002/14651858.CD011300.pub3. PMID 34870327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent, Step 2 [randomized part]): 03 Feb 2010/15 Feb 2012. Clinical data cut-off: 01 May 2014. Study completion date: 15 June 2015
Pre-assignment Details: Enrolled: 197 screened for eligibility; 25 excluded (mainly due to non-fulfillment of inclusion or exclusion criteria) and 172 subjects randomized.
Groups:
- Tecemotide (L-BLP25) + Cyclophosphamide: Single dose of cyclophosphamide (300 milligrams per square meter [mg/m^2] to a maximum of 600 mg) was administered intravenously, 3 days prior to the start of vaccination, followed by weekly subcutaneous vaccinations with tecemotide (L-BLP25) (930 microgram [mcg]) for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with tecemotide (L-BLP25) (930 mcg) were administered every 6 weeks until progressive disease (PD) was documented.
- Placebo + Saline: Single dose of saline (sodium chloride, 9 grams per liter [g/L]) was administered intravenously, 3 days prior to the start of vaccination, followed by weekly subcutaneous vaccinations with placebo doses matched to tecemotide (L-BLP25) for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with placebo were administered every 6 weeks until PD was documented.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Started | 114 | 58
Completed | 95 | 43
Not Completed | 19 | 15
Not completed — Ongoing treatment at data cut-off date | 19 | 15

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) analysis set included all subjects randomly allocated to a treatment (tecemotide [L-BLP25] or placebo)
Groups:
- Tecemotide (L-BLP25) + Cyclophosphamide: Single dose of cyclophosphamide (300 milligrams per square meter [mg/m^2] to a maximum of 600 mg) was administered intravenously, 3 days prior to the start of vaccination, followed by weekly subcutaneous vaccinations with tecemotide (L-BLP25) (930 mcg) for 8 weeks, followed by a maintenance treatment phase starting at Week 14, in which subcutaneous vaccinations with tecemotide (L-BLP25) (930 mcg) were administered every 6 weeks until PD was documented.
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline | Total
Number analyzed (Participants) | 114 | 58 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.31) | 60.1 (9.81) | 62.0 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 98 | 47 | 145

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: OS time was defined as the time from randomization to death. Participants without event were censored at the last date known to be alive or at the clinical cut-off date (01 May 2014), whichever was earlier.
Time Frame: Time from randomization to death or last day known to be alive reported between day of first subject randomized in Step 2 (i.e. 03 Feb 2010), until clinical cut-off date (i.e. 01 May 2014).
Population: ITT analysis set included all subjects randomly allocated to a treatment (tecemotide [L-BLP25] or placebo).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 114 | 58
Months | 32.4 [26.7 to NA] — Since there were not enough participants with an event, the upper limit was not estimable. | 32.2 [19.6 to NA] — Since there were not enough participants with an event, the upper limit was not estimable.
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) + Cyclophosphamide vs Placebo + Saline; Test type: Superiority or Other; p = 0.828, Log Rank — This trial was not powered to demonstrate statistical significance of treatment differences with respect to a statistical test, i.e., the p value being lower than a significance level of alpha (α) = 0.05; Hazard Ratio (HR) = 0.953, 95% CI 2-sided [0.614 to 1.479] — Cox proportional hazards regression model

2. Secondary Outcome: Time To Progression (TTP) - Investigator Read
Description: TTP was defined as the time from date of randomization to date of radiological diagnosis of PD (based on Response Evaluation Criteria in Solid Tumors [RECIST] v1.0). In the event that radiological confirmation could not be obtained but participant was withdrawn from trial treatment or died due to disease progression, TTP was measured from date of randomization to the date of discontinuation of trial treatment. Participants without event who died from causes other than disease progression were censored at date of death. Participants without event who were lost to follow-up were censored at the date of lost to follow-up, except if they missed 2 consecutive scheduled doses, in which case they were considered as having disease progression at time of first missed administration. Participants without event with ongoing treatment at time of analysis, or who had stopped treatment for reasons other than PD, were censored on the date of last treatment administration.
Time Frame: Time from randomization to PD, reported between day of first subject randomized in Step 2 (i.e. 03 Feb 2010), until clinical cut-off date (i.e. 01 May 2014).
Population: ITT Analysis Set included all subjects randomly allocated to a treatment (tecemotide [L-BLP25] or placebo).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 114 | 58
Months | 11.3 [6.5 to 12.9] | 7.0 [5.8 to 14.2]

3. Secondary Outcome: Progression Free Survival (PFS) Time - Investigator Read
Description: PFS time was defined as the duration from randomization to either first observation of objective PD (based on RECIST v1.0) or occurrence of death due to any cause. Participants without event still on treatment at time of analysis, or who stopped treatment for reasons other than PD or PD without radiological confirmed progression, were censored at the last imaging date. Participants without event who were lost to follow-up were censored at the date of lost to follow-up, except if they missed 2 consecutive scheduled doses, in which case they were considered as having disease progression at time of first missed administration.
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first subject randomized in Step 2 (i.e. 03 Feb 2010), until clinical cut-off date (i.e. 01 May 2014).
Population: ITT analysis set included all subjects randomly allocated to a treatment (tecemotide [L-BLP25] or placebo).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 114 | 58
Months | 11.6 [6.9 to 13.9] | 8.0 [5.9 to 14.2]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the duration from date of randomization to the date of discontinuation of any trial treatment (cyclophosphamide or saline, tecemotide [L-BLP25] or placebo vaccine) for any reason as reported by the Investigator. Participants who had missed 2 consecutive scheduled doses and were subsequently lost to follow-up were considered as treatment failures with event date as date of first missed administration. Participants without event still on treatment at time of analysis were censored on the date of last treatment administration.
Time Frame: Time from randomization to discontinuation of trial treatment, reported between day of first subject randomized in Step 2 (i.e. 03 Feb 2010), until clinical cut-off date (i.e. 01 May 2014).
Population: ITT analysis set included all subjects randomly allocated to a treatment (tecemotide [L-BLP25] or placebo).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Number analyzed (Participants) | 114 | 58
Months | 8.0 [4.6 to 11.5] | 6.2 [3.2 to 11.5]

ADVERSE EVENTS:
Time Frame: Time from first dosing day of trial treatment until 42 days after last dose of trial treatment or the clinical data cut-off date (01 May 2014).
Description: Safety analysis set included all subjects who were treated with tecemotide [L-BLP25] or placebo. Reported treatment-emergent adverse events included events that emerged during treatment having been absent pre-treatment, or worsened relative to the pre-treatment state.
Arm/Group | Tecemotide (L-BLP25) + Cyclophosphamide | Placebo + Saline
Serious Adverse Events (participants affected / at risk) | 24/114 | 12/57
Other Adverse Events (participants affected / at risk) | 107/114 | 53/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=114) | Placebo + Saline (N=57)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Gingival cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecemotide (L-BLP25) + Cyclophosphamide (N=114) | Placebo + Saline (N=57)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 12 (12) | 2 (2)
Dental caries (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 5 (5)
Nausea (Gastrointestinal disorders) | 13 (13) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 7 (7) | 6 (6)
Influenza like illness (General disorders) | 7 (7) | 3 (3)
Injection site erythema (General disorders) | 10 (10) | 1 (1)
Injection site nodule (General disorders) | 9 (9) | 0 (0)
Malaise (General disorders) | 8 (8) | 5 (5)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 9 (9) | 2 (2)
Herpes zoster (Infections and infestations) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 33 (33) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 36 (36) | 14 (14)
Weight increased (Investigations) | 7 (7) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)
Hypertension (Vascular disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other